CLINICAL TRIAL: NCT05365542
Title: Mapping of Anticoagulation in Chronic Hemodialysis Patients Versus Hemodialyzer Fiber Patency, Bleedings and Quality of Life
Brief Title: Anticoagulation in Chronic Hemodialysis Patients Versus Hemodialyzer Fiber Patency, Bleedings and Quality of Life
Acronym: ClotSigns
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: UGent_ClotSigns
Record Dates: First submitted 2022-01-19; First posted 2022-05-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Blood Coagulation
Keywords: Hemodialyzer; Fibre Clotting; Quality of life; Bleeding; Bruising
MeSH Terms: conditions — Thrombosis; Hemorrhage; Contusions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hemodialyzer scanning — After the hemodialysis session, the used dialyzer is rinsed and dried before scanning in a Micro Computed Tomography scanner. From cross-sectional images, the number of patent fibers is quantified.
Other: Bleeding Questionnaires — The ISTH Bleeding Assessment Tool and the HASBLED questionnaires are asked
Other: Quality of life questionnaire — The EQ5D questionnaire is asked.
Other: Visual inspection of the limbs — Visual inspection is done of the patient's limbs in order to quantify bruising.

SUMMARY:
Stable chronic hemodialysis patients are included in this observational study. After a midweek dialysis (test moment 1), the hemodialyzer is dried and scanned in a micro Computed Tomography scanner to quantify the number of patent fibers. All dialysis parameters are collected as well as the anticoagulation dose. During the same session, patients are asked about their bleeding and quality of life status. Four (test moment 2) respectively eight weeks later (test moment 3), patients are asked again for their bleeding and quality of life status using validated questionnaires.

DETAILED DESCRIPTION:
All stable chronic hemodialysis (HD) patients having daytime dialysis in the Ghent University Hospital, are included.

From the patient's record, data are collected: demographic data (i.e. age, weight, dialysis vintage), blood data related to clotting (i.e. number of platelets, hemoglobin, International Normalized Ratio (INR), C-reactive protein (CRP)). All data is pseudomized.

The study has three test moments. During the entire study, patients are dialyzed with their usual dialyzer on their usual dialysis machine and with their usual dialysis settings and anticoagulation dosis. After the first midweek test session (test moment 1), the used hemodialyzer is rinsed with the standard rinsing procedure, dried in blood and dialysate compartment with positive pressure ventilation during 12-24h, eventually stored at 5°C, and finally scanned in a micro-CT scan in order to quantify the number of patent fibers. The dialyzer is vertically mounted on a rotating disc in front of the X-ray bundle. Scans are made every 0.15° with 2401 projections during 500ms each. After image reconstruction, visualisation are obtained from cross-sections of the hemodialyzer. Open fibers are counted with an open source computer program used for biological image analysis. By comparing the number of open fibers with the total number of fibers in an unused hemodialyzer, the percentage of open fibers can be quantified.

During the same week of the first test moment, several validated questionnaires will be completed: questionnaires about intention for bleeding (i.e. the International Society of Thrombosis and Haemostasis (ISHT) Bleeding Assessment Tool and the Hypertension, Abnormal Renal/Liver Function, Stroke, Bleeding History or Predisposition, Labile INR, Elderly, Drugs/Alcohol Concomitantly (HASBLED) score), and a questionnaire about quality of life (i.e. EuroQoL 5D (EQ5D)). Besides, a visual inspection is performed of the limbs of the patient in order to quantify bruising.

By comparing the percentage of open fibers with the administered anticoagulation dosis and the different questionnaires about bleeding, mutual relations can be drawn.

In order to check reliability, questionnaires and visual inspection are repeated after 4 weeks and 8 weeks (test moments 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* treated with chronic daytime hemodialysis

Exclusion Criteria:

* no active infection at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable chronic hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Relation between anticoagulation dose and number of patent dialyzer fibers | 8 weeks
  By comparing the anticoagulation dose with the number of patent fibers as measured post dialysis by visualising the dialyzer in a micro computed tomography (CT) machine and by counting the number of open fibers in a cross-section at the dialyzer outlet.
Relation between anticoagulation dose and bleeding score | 8 weeks
  Two validated questionnaires about bleeding are used: International Society on Thrombosis and Hemostasis Bleeding Assessment Tool (ISTH BAT) and the Hypertension, Abnormal Renal/Liver Function, Stroke, Bleeding History or Predisposition, Labile INR, Elderly, Drugs/Alcohol (HASBLED). ISTH BAT score can be 0-56, with a score >4 (male) and >6 (female) to be considered as abnormal. HASBLED score can be 0-9 with a score >2 to be considered as a patient with high risk of bleeding.
  Scores are related to the administered anticoagulation dose.
Relation between bleeding score and quality of life score | 8 weeks
  Scores of the validated questionnaires about bleeding are related to the EuroQol Five Dimensions questionnaire (EQ5D) about quality of life. Scores per question are 1 to 3. Analysis is done with an online system accounting for patient's age.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, Principal Investigator — UZ Gent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided